CLINICAL TRIAL: NCT03024840
Title: The Effect of Sevoflurane or Propofol on Brain Injury and Neurocognitive in Pediatric Living Related Liver Transplantation
Brief Title: Anaesthetic and Pediatric Living Related Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tianjin First Central Hospital (Other)
Responsible Party: Principal Investigator, Wenli Yu, Wenli Yu,PhD ,Department of Anesthesiology,Tianjin First Center Hospital, Tianjin First Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016N0039KY
Record Dates: First submitted 2016-12-23; First posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Liver Transplantation; Children
Keywords: Propofol; Neurocognitive Disorders; Liver transplantation; Pediatrics; Brain Injuries
MeSH Terms: conditions — Neurocognitive Disorders; Brain Injuries | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sevoflurane (Experimental): Sevoflurane is inhalated with 1%-2% after anesthesia induction until end of the surgery.
  Interventions: Drug: Sevoflurane
- propofol (Experimental): Propofol is injected with 9-15 mg/kg/h after anesthesia induction until end of the surgery.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane: 1%~2%
  Arms: sevoflurane
Drug: Propofol — Propofol: 9-15 mg/kg/h
  Arms: propofol

SUMMARY:
To study the effect of different anaesthetic methods on pediatric neurocognitive development and cerebral injury during pediatric living related liver transplantation .

DETAILED DESCRIPTION:
Since the 1960 s, with the successful development of liver transplantation, it has become an important method for the treatment of patients with end-stage liver disease.Biliary atresia1 is the most frequent causes of pediatric end-stage liver disease,.The morbidity of congenital biliary atresia is 1/8000-18, 0002 ,which influence the patients' overall growth and development situation. The rising of living donor liver transplantation has provide children with the chance of a timely treatment since the 1980 s, It is no doubt that pediatric liver transplantation is facing with many complications, including the most importance of neurocognitive development .Now the researches of neurological complications is less .According to statistics, the incidence of neurological complications after pediatric liver transplantation was 8% - 46% . So it is necessary to research the neurological complications and brain protection strategy .Previous studies have studied that some anaesthetic have uncertain affect on the development of children.

ELIGIBILITY:
Inclusion Criteria:

* Children with end-stage liver disease Children with biliary atresia

Exclusion Criteria:

* pre-existing cerebral disease second liver transplantation

Ages: 4 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evidence of cerebral injury including S-100 β protein, neurospecific enolase confirmed by electrochemiluminescence | before skin incision, 0.5 hour after anhepatic,1 hour of neohepatic stage,the end of surgery,24 hours after operation
Evidences of inflammatory factor such as interleukin-6，interleukin-10，et al confirmed by electrochemiluminescence | before skin incision, 0.5 hour after anhepatic,1 hour of neohepatic stage,the end of surgery,24 hours after operation

SECONDARY OUTCOMES:
Evaluation of neurocognitive disorder using Bayley Scales of Infant Development | 1 day before surgery, 7days,14 days and 21days of post-operation
Evaluation of delirium using Pediatric Anesthesia Emergence Delirium | Within 1 days after extubation
hemodynamics index | before skin incision, 0.5 hour after anhepatic,1 hour of neohepatic stage,the end of surgery,24 hours after operation

CONTACTS AND LOCATIONS:
Locations (1):
- No.24 Fukang Road,Nankai District, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No